CLINICAL TRIAL: NCT01959126
Title: The Effect of a Stress Reduction Program Using Mindfulness Techniques on Markers of Cellular Stress and Aging
Brief Title: Health Enhancement And Resilience Training
Acronym: HEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10-02063
Record Dates: First submitted 2013-07-10; First posted 2013-10-09 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Stress; Aging; Well-being
Keywords: Telomerase; Telomere length; Psychological Sress; Mindfulness
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stress-reduction class (Experimental): Study participants enrolled in a 12-week stress reduction course based on the principles of mindfulness. They attended four six-hour workshops and participated in 12 weekly hour-long web video conferencing calls to reinforce what was taught in the workshops. We have two groups: chronically-stressed maternal caregivers of children on the autism spectrum and control mothers whose children have no significant psychiatric or physical impairment.
  Interventions: Behavioral: Stress-reduction class

INTERVENTIONS:
Behavioral: Stress-reduction class — Study participants enrolled in a 12-week stress reduction course based on the principles of mindfulness. They attended four six-hour workshops and participated in 12 weekly hour-long web video conferencing calls to reinforce what was taught in the workshops. We have two groups: chronically-stressed maternal caregivers of children on the autism spectrum and control mothers whose children have no significant psychiatric or physical impairment. Both groups received similar instruction.
  Other Names: mindfulness

SUMMARY:
The purpose of this research study is to examine whether a stress reduction intervention can improve health, mood and biological markers of cellular stress and aging in a group of chronically-stressed maternal caregivers and healthy maternal controls.

DETAILED DESCRIPTION:
This stress-reduction intervention was added into an ongoing observational study in May of 2013. The parent study is a prospective cohort study of the effects of chronic stress in a group of maternal caregivers with children on the autism spectrum and healthy controls whose children have no diagnosis. Study participants are being invited to enroll in a 12-week stress reduction course based on the principles of mindfulness. They will attend four six-hour workshops and participate in 12 weekly hour-long web video conferencing calls to reinforce what is taught in the workshops.

At the beginning and the end of the intervention, they complete self-report measures of psychological well-being and give saliva samples. Since the women are also participating in the longitudinal study, we have other before and after data for them. These include psycho-social measures, body measurements, psycho-physiology measurements, cognitive tests, actigraphy (for sleep), as well as saliva (for hormones), hair (for hormones) and blood (for telomeres, telomerase, gene expression, circulating hormones, inflammation and oxidative stress).

ELIGIBILITY:
Inclusion Criteria:

* Must have at least one child between 2 and 16 at time of enrollment
* Caregivers must have a child diagnosed in that age range diagnosed with an autism spectrum disorder.
* Controls must have a healthy child in that age range. All women must be

Exclusion Criteria:

* Chronic disease, including recent history of cancer
* History of psychiatric disorder, such as bipolar disorder or post-traumatic stress disorder
* Medications, including statins, anti-anxiety drugs, and for controls only anti-depressants.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Salivary telomere length | Change from beginning to end of 12-week intervention
  Participants will give saliva samples at the beginning and the end of the intervention. Salivary telomere length will be analyzed at both time points.

SECONDARY OUTCOMES:
Psychological Well-Being | Change from beginning to end of 12-week intervention
  We will collect perceived stress, acceptance and awareness of emotions and rumination at the beginning and at the end of the intervention.
Telomere length from blood cells | Change over six months pre- and post-intervention
  Since participants are also taking part in an ongoing non-interventional longitudinal study, they will provide blood samples at their 18-month study visit, which occurs before the start of the intervention, and at the 24-month study visit, which occurs after the end of the intervention. We will measure telomere length pre- and post-intervention in a variety of blood cell types.
Telomerase | Change over 6 months pre- and post-intervention
  Since participants are also taking part in an ongoing non-interventional longitudinal study, they will provide blood samples at their 18-month study visit, which occurs before the start of the intervention, and at the 24-month study visit, which occurs after the end of the intervention. We will measure telomerase pre- and post-intervention in a variety of blood cell types.
Cognitive functioning | Change over six months pre- and post-intervention
  Since participants are also taking part in an ongoing non-interventional longitudinal study, they will complete a battery of cognitive tasks at their 18-month study visit, which occurs before the start of the intervention, and at the 24-month study visit, which occurs after the end of the intervention. We will be able to assess performance pre- and post-intervention, to see if it improves after the stress-reduction training.

CONTACTS AND LOCATIONS:
Overall Officials: Elissa S Epel, PhD, Principal Investigator — University of California, San Francisco; Elizabeth Blackburn, PhD, Principal Investigator — University of California, San Francisco; Jue Lin, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States